CLINICAL TRIAL: NCT07164365
Title: Decisional Conflict in Patients With Advanced Cancer in a Shared Decision-Making Model: A Randomized Clinical Trial
Brief Title: Effect of an Interdisciplinary Shared Decision-Making Intervention on Decisional Conflict in Advanced Cancer Patients Receiving Third-Line Therapy
Acronym: SharedDecision
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-CIE-0357-25; FM-CIE-0357-25 (Other: Hospital Universitario San Ignacio)
Record Dates: First submitted 2025-07-28; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Decisional Conflict, Advanced/Metastatic Solid Tumors, Shared Decision-making
Keywords: Cancer, advanced disease, decisional conflict, shared decision making, interdisciplinary intervention, oncology, palliative care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial; parallel two-arm design (intervention and control)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm: Interdisciplinary shared decision-making consultation (Active Comparator): Interdisciplinary shared decision-making consultation (with oncologist, palliative care physician, psychologist) following a six-step shared decision-making process.
  Interventions: Behavioral: Interdisciplinary Shared Decision-Making Consultation
- Control arm (No Intervention): Standard oncology consultation

INTERVENTIONS:
Behavioral: Interdisciplinary Shared Decision-Making Consultation — One additional face-to-face consultation with a team (oncologist, palliative care, psychologist), following a six-step shared decision-making process.
  Arms: Intervention Arm: Interdisciplinary shared decision-making consultation

SUMMARY:
The study aims to evaluate whether an interdisciplinary intervention based on a shared decision-making model can reduce decisional conflict in patients with metastatic solid tumors (lung, breast, colorectal, prostate, or ovarian cancer) who are indicated for third-line systemic treatment. Participants are randomized to receive either standard oncology consultation or an additional interdisciplinary consultation involving oncology, palliative care, and psychology. The intervention emphasizes providing information and support for treatment decisions.

DETAILED DESCRIPTION:
* Problem Statement: In Colombia, advanced cancer is common and treatment options become increasingly complex by the third line of therapy, often lacking standardized guidelines. This complexity, along with uncertainty about prognosis and treatment benefits, can lead to significant decisional conflict for patients.
* Objective: To determine whether a structured interdisciplinary intervention using shared decision-making reduces decisional conflict compared to standard care.
* Population: Adults (≥18 years) with metastatic lung, breast, colon, ovary, or prostate cancer at Hospital San Ignacio, eligible for third-line systemic therapy.
* Intervention: The intervention group receives an additional consultation involving a medical oncologist, palliative care physician, and psychologist. The session follows six steps: inviting the patient to participate, describing options, detailing benefits and risks, clarifying patient goals, facilitating decision deliberation, and outlining next steps-all based on the shared decision-making model.
* Control Group: Receives standard oncology consultation only.
* Randomization: Assignment is done randomly and independently.
* Outcomes:
* Primary: Decisional conflict measured by the Decisional Conflict Scale.
* Secondary: Patient satisfaction, decision regret, perceptions of shared decision-making, symptom burden, and levels of neuroticism, all assessed with validated instruments.
* Sample Size: 62 participants (31 per group) are planned, allowing for potential losses.
* Follow-up: Patients are assessed immediately after intervention/consultation and again at three months.
* Analysis: Data will be analyzed by intention-to-treat, using quantitative scales, and adjusting for confounding factors. Subgroup analyses by demographic and clinical characteristics are planned.

Overall, the study is designed to inform best practices on supporting advanced cancer patients in complex treatment decisions, exploring the effects of an interdisciplinary, patient-centered intervention on decisional conflict and related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Diagnosed with metastatic lung, breast, colon, ovary, or prostate cancer
* Have completed two prior lines of systemic therapy
* Indication for third-line systemic therapy (chemotherapy, immunotherapy, or hormone therapy)
* Under follow-up at Hospital San Ignacio
* Capacity to provide informed consent
* Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2025-08-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Score | Immediately post-intervention
  Measured using the Decisional Conflict Scale (16 items); score ≥25 defines clinically significant conflict

SECONDARY OUTCOMES:
Patient satisfaction | Immediately post-intervention and at 3 months follow-up
  Measure of the importance of patient satisfaction as a key quality indicator and highlights the use of the Likert scale as an effective tool for measuring perceptions of healthcare quality. The objective is to evaluate patient satisfaction by using the Likert scale, where scores of 7 denote satisfaction, and scores different from 7 indicate dissatisfaction.
Decision regret | at 3 months after de intervention
  Use of the Decision Regret Scale (EAD) to measure patients' regret after making healthcare decisions. The objective is to assess the level of decision regret, with higher scores indicating greater regret, to better understand patients' emotional responses and improve decision-making processes.
Perspective on shared decision-making | Immediately post-intervention
  This is a short, patient-centered questionnaire to assess the shared decision-making process in clinical settings. It is psychometrically robust, easy to use, and provides both an overall score and item-level insights, making it valuable for evaluating interventions and improving patient-physician collaboration in healthcare decisions.
Symptom burden | 1 day after intervention and 3 months post intervention
  We are going to measure this using the Edmonton Symptom Assessment Scale (ESAS) is a brief, patient-completed tool designed to assess the severity of common symptoms in palliative care, especially among cancer patients. It uses 10 visual numeric scales to evaluate both physical and psychological symptoms, is validated in multiple languages, and is widely used in clinical and research settings for ongoing symptom monitoring.
Neuroticism trait | Immediately post-intervention
  We are going to measure this using the MMPI-2, which is a comprehensive psychological assessment tool designed to evaluate a wide range of personality traits and psychopathological conditions. It is widely used in clinical and research settings, and for this study, only the neuroticism dimension will be assessed using a subset of 33 items. The results are interpreted using standardized T scores, with higher scores indicating greater psychological distress or maladaptive traits.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario San Ignacio, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Yes
We will share the demographic data of the participants in our database.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Ministerio de salud. Resolución 8430 de 1993. 1993. p. 1-19
- [Background] Ben-Porath YS, Hosteller K, Butcher JN, Graham JR, Ben-Porath S. New Subscales for the MMPI-2 Social Introversion (Si) Scale. Vol. l, Psychological Assessment: A Journal of Consulting and Clinical Psychology. 1989
- [Background] Jiménez OR. Interpretación clínica y psicodinámica del MMP1: inventario multifásico de la personalidad de Minnesota. Diana. 1987;
- [Background] Trull TJ, David Useda J, Costa PT, Mccrae RR. Comparison of the MMPI-2 Personality Psychopathology Five (PSY-5), the NEO-PI, and the NEO-PI-R. Psychological Assessment. 1995
- [Background] Harkness AR, Mcnulty JL, Ben-Porath YS. The Personality Psychopathology Five (PSY-5) : Constructs and MMPI-2 Scales. Vol. 7, Psychological Assessment. 1995
- [Background] Gordon RM, Stoffey RW, Perkins BL. Comparing the Sensitivity of the MMPI-2 Clinical Scales and the MMPI-RC Scales to Clients Rated as Psychotic, Borderline or Neurotic on the Psychodiagnostic Chart. Psychology. 2013;04(09):12-6.
- [Background] Butcher JN, Graham JR, Ben-Porath YS, Tellegen A, Dahlstrom WG, Kaemmer B, et al. MMPI®-2 Inventario Multifásico de Personalidad de Minnesota®-2 Comité de tipificación del MMPI ®-2: Adaptación española: Manual. 2019
- [Background] Carvajal A, Centeno C, Watson R, Bruera E. A comprehensive study of psychometric properties of the Edmonton Symptom Assessment System (ESAS) in Spanish advanced cancer patients. Eur J Cancer. 2011 Aug;47(12):1863-72. doi: 10.1016/j.ejca.2011.03.027. Epub 2011 Apr 22. PMID 21514818
- [Background] Aktas A, Walsh D, Kirkova J. The psychometric properties of cancer multisymptom assessment instruments: a clinical review. Support Care Cancer. 2015 Jul;23(7):2189-202. doi: 10.1007/s00520-015-2732-7. Epub 2015 Apr 19. PMID 25894883
- [Background] Nekolaichuk C, Watanabe S, Beaumont C. The Edmonton Symptom Assessment System: a 15-year retrospective review of validation studies (1991--2006). Palliat Med. 2008 Mar;22(2):111-22. doi: 10.1177/0269216307087659. PMID 18372376
- [Background] Chang VT, Hwang SS, Feuerman M. Validation of the Edmonton Symptom Assessment Scale. Cancer. 2000 May 1;88(9):2164-71. doi: 10.1002/(sici)1097-0142(20000501)88:93.0.co;2-5. PMID 10813730
- [Background] Llanos Zavalaga F, Rosas Aguirre A, Mendoza Requena D, Contreras Ríos C. Universidad Peruana Cayetano Heredia. Rev Med Hered. 2001;12(2):52-7
- [Background] Floriano N, Aranda R, Manuel J, González R, Maribel A, Rodríguez A, et al. Validación de Shared Decision Making Questionnaire-physician version (SDM-Q-Doc) en español Revista Clínica de. Medicina de Familia (Internet). 2020;13(3):190-7. Available from: http://www.redalyc.org/articulo.oa?id=169664978003
- [Background] De las Cuevas C, Perestelo-Perez L, Rivero-Santana A, Cebolla-Marti A, Scholl I, Harter M. Validation of the Spanish version of the 9-item Shared Decision-Making Questionnaire. Health Expect. 2015 Dec;18(6):2143-53. doi: 10.1111/hex.12183. Epub 2014 Mar 5. PMID 24593044
- [Background] Charles C, Gafni A, Whelan T. Decision-making in the physician-patient encounter: revisiting the shared treatment decision-making model. Soc Sci Med. 1999 Sep;49(5):651-61. doi: 10.1016/s0277-9536(99)00145-8. PMID 10452420
- [Background] Urrutia M, Campos S, O'Connor A. [Validation of a Spanish version of the Decisional Conflict scale]. Rev Med Chil. 2008 Nov;136(11):1439-47. doi: 10.4067/s0034-98872008001100010. Spanish. PMID 19301775
- [Background] Wang MM, Loh EW, Chou JF, Sung PM, Chou YY, Lin YK, Chen SF, Tam KW. Influence of Shared Decision Making on Decisional Conflict and Regret in Postpartum Mother-Infant Care: A Randomized Controlled Trial. Value Health. 2021 Sep;24(9):1335-1342. doi: 10.1016/j.jval.2021.03.011. Epub 2021 May 3. PMID 34452714
- [Background] Niburski K, Guadagno E, Abbasgholizadeh-Rahimi S, Poenaru D. Shared Decision Making in Surgery: A Meta-Analysis of Existing Literature. Patient. 2020 Dec;13(6):667-681. doi: 10.1007/s40271-020-00443-6. PMID 32880820
- [Background] Levy D, Dhillon HM, Lomax A, Marthick M, McNeil C, Kao S, Lacey J. Certainty within uncertainty: a qualitative study of the experience of metastatic melanoma patients undergoing pembrolizumab immunotherapy. Support Care Cancer. 2019 May;27(5):1845-1852. doi: 10.1007/s00520-018-4443-3. Epub 2018 Sep 4. PMID 30178142
- [Background] Roccas S, Sagiv L, Schwartz SH, Knafo A. The Big Five personality factors and personal values. Pers Soc Psychol Bull. 2002;28(6):789-801
- [Background] Komarraju M, Karau SJ, Schmeck RR, Avdic A. The Big Five personality traits, learning styles, and academic achievement. Pers Individ Dif. 2011 Sep;51(4):472-7
- [Background] Di Fabio A, Saklofske DH, Gori A, Svicher A. Perfectionism: A network analysis of relationships between the Big Three Perfectionism dimensions and the Big Five Personality traits. Pers Individ Dif. 2022 Dec 1;199
- [Background] Markon KE. Hierarchies in the Structure of Personality Traits. Soc Personal Psychol Compass. 2009 Sep;3(5):812-26
- [Background] Zuckerman M, Kuhlman DM, Joireman J, Teta P, Kraft M. A Comparison of Three Structural Models for Personality: The Big Three, the Big Five, and the Alternative Five. Vol. 65, Journal of Personality and Social Psychology. 1993
- [Background] Barlow DH, Ellard KK, Sauer-Zavala S, Bullis JR, Carl JR. The Origins of Neuroticism. Perspect Psychol Sci. 2014 Sep;9(5):481-96. doi: 10.1177/1745691614544528. PMID 26186755
- [Background] Roemer L, Salters K, Raffa SD, Orsillo SM. Fear and avoidance of internal experiences in GAD: Preliminary tests of a conceptual model. Vol. 29, Cognitive Therapy and Research. 2005. p. 71-88
- [Background] McLaughlin KA, Mennin DS, Farach FJ. The contributory role of worry in emotion generation and dysregulation in generalized anxiety disorder. Behav Res Ther. 2007 Aug;45(8):1735-52. doi: 10.1016/j.brat.2006.12.004. Epub 2006 Dec 28. PMID 17270145
- [Background] Watson D, Clark LA, Harkness AR. Structures of personality and their relevance to psychopathology. J Abnorm Psychol. 1994 Feb;103(1):18-31. PMID 8040477
- [Background] McCrae RR, Costa PT. Personality in adulthood: A five- factor theory perspective. . 2nd ed. New York: Guilford Press; 2003
- [Background] Weiss A, Costa PT Jr. Domain and facet personality predictors of all-cause mortality among Medicare patients aged 65 to 100. Psychosom Med. 2005 Sep-Oct;67(5):724-33. doi: 10.1097/01.psy.0000181272.58103.18. PMID 16204430
- [Background] Kates JM. Treatment-related Decisional Conflict, Quality of Life, and Comorbidity in Older Adults with Cancer. Asia Pac J Oncol Nurs. 2018 Oct-Dec;5(4):421-429. doi: 10.4103/apjon.apjon_32_18. PMID 30271826
- [Background] Baek SK, Kim SY, Heo DS, Yun YH, Lee MK. Effect of advanced cancer patients' awareness of disease status on treatment decisional conflicts and satisfaction during palliative chemotherapy: a Korean prospective cohort study. Support Care Cancer. 2012 Jun;20(6):1309-16. doi: 10.1007/s00520-011-1218-5. Epub 2011 Jul 1. PMID 21720748
- [Background] Baca-Dietz D, Wojnar DM, Espina CR. The shared decision-making model: Providers' and patients' knowledge and understanding in clinical practice. J Am Assoc Nurse Pract. 2020 Jun 30;33(7):529-536. doi: 10.1097/JXX.0000000000000401. PMID 32618736
- [Background] Arch JJ, Bright EE, Finkelstein LB, Fink RM, Mitchell JL, Andorsky DJ, Kutner JS. Anxiety and Depression in Metastatic Cancer: A Critical Review of Negative Impacts on Advance Care Planning and End-of-Life Decision Making With Practical Recommendations. JCO Oncol Pract. 2023 Dec;19(12):1097-1108. doi: 10.1200/OP.23.00287. Epub 2023 Oct 13. PMID 37831973
- [Background] Ter Stege JA, Oldenburg HSA, Woerdeman LAE, Witkamp AJ, Kieffer JM, van Huizum MA, van Duijnhoven FH, Hahn DEE, Gerritsma MA, Kuenen MA, Kimmings NAN, Ruhe QPQ, Krabbe-Timmerman IS, Riet MV, Corten EML, Sherman KA, Bleiker EMA. Decisional conflict in breast cancer patients considering immediate breast reconstruction. Breast. 2021 Feb;55:91-97. doi: 10.1016/j.breast.2020.12.001. Epub 2020 Dec 9. PMID 33387811
- [Background] Calderon C, Ferrando PJ, Lorenzo-Seva U, Higuera O, Ramon Y Cajal T, Rogado J, Mut-Lloret M, Rodriguez-Capote A, Jara C, Jimenez-Fonseca P. Validity and Reliability of the Decision Regret Scale in Cancer Patients Receiving Adjuvant Chemotherapy. J Pain Symptom Manage. 2019 Apr;57(4):828-834. doi: 10.1016/j.jpainsymman.2018.11.017. Epub 2019 Jan 11. PMID 30639730
- [Background] Gilovich T, Medvec VH. The experience of regret: what, when, and why. Psychol Rev. 1995 Apr;102(2):379-95. doi: 10.1037/0033-295x.102.2.379. PMID 7740094
- [Background] Hotta K, Kiura K, Takigawa N, Yoshioka H, Hayashi H, Fukuyama H, Nishiyama A, Yokoyama T, Kuyama S, Umemura S, Kato Y, Nogami N, Segawa Y, Yasugi M, Tabata M, Tanimoto M. Desire for information and involvement in treatment decisions: lung cancer patients' preferences and their physicians' perceptions: results from Okayama Lung Cancer Study Group Trial 0705. J Thorac Oncol. 2010 Oct;5(10):1668-72. doi: 10.1097/JTO.0b013e3181f1c8cb. PMID 20871267
- [Background] Mallinger JB, Shields CG, Griggs JJ, Roscoe JA, Morrow GR, Rosenbluth RJ, Lord RS, Gross H. Stability of decisional role preference over the course of cancer therapy. Psychooncology. 2006 Apr;15(4):297-305. doi: 10.1002/pon.954. PMID 16041829
- [Background] Ankolekar A, De Ruysscher D, Reymen B, Houben R, Dekker A, Roumen C, Fijten R. Shared decision-making for prophylactic cranial irradiation in extensive-stage small-cell lung cancer: an exploratory study. Transl Lung Cancer Res. 2021 Jul;10(7):3120-3131. doi: 10.21037/tlcr-21-175. PMID 34430352
- [Background] Pecanac KE, Brown RL, Steingrub J, Anderson W, Matthay MA, White DB. A psychometric study of the decisional conflict scale in surrogate decision makers. Patient Educ Couns. 2018 Nov;101(11):1957-1965. doi: 10.1016/j.pec.2018.07.006. Epub 2018 Jul 7. PMID 30054105
- [Background] Coronado-Vazquez V, Canet-Fajas C, Delgado-Marroquin MT, Magallon-Botaya R, Romero-Martin M, Gomez-Salgado J. Interventions to facilitate shared decision-making using decision aids with patients in Primary Health Care: A systematic review. Medicine (Baltimore). 2020 Aug 7;99(32):e21389. doi: 10.1097/MD.0000000000021389. PMID 32769870
- [Background] Jeon BM, Kim SH, Lee SJ. Decisional conflict in end-of-life cancer treatment among family surrogates: A cross-sectional survey. Nurs Health Sci. 2018 Dec;20(4):472-478. doi: 10.1111/nhs.12537. Epub 2018 Jun 19. PMID 29920890
- [Background] Lenz ER, Pugh LC. Middle range theory for nursing. 3rd ed. Smith Mary Jane, Liehr Patricia R., editors. NewYork: Springer; 2014. 95-165 p
- [Background] Emanuel EJ, Emanuel LL. Four models of the physician-patient relationship. JAMA. 1992 Apr 22-29;267(16):2221-6. No abstract available. PMID 1556799
- [Background] Kane HL, Halpern MT, Squiers LB, Treiman KA, McCormack LA. Implementing and evaluating shared decision making in oncology practice. CA Cancer J Clin. 2014 Nov-Dec;64(6):377-88. doi: 10.3322/caac.21245. Epub 2014 Sep 8. PMID 25200391
- [Background] Laidsaar-Powell R, Butow P, Bu S, Charles C, Gafni A, Fisher A, Juraskova I. Family involvement in cancer treatment decision-making: A qualitative study of patient, family, and clinician attitudes and experiences. Patient Educ Couns. 2016 Jul;99(7):1146-1155. doi: 10.1016/j.pec.2016.01.014. Epub 2016 Jan 28. PMID 26873544
- [Background] Gennari A, Andre F, Barrios CH, Cortes J, de Azambuja E, DeMichele A, Dent R, Fenlon D, Gligorov J, Hurvitz SA, Im SA, Krug D, Kunz WG, Loi S, Penault-Llorca F, Ricke J, Robson M, Rugo HS, Saura C, Schmid P, Singer CF, Spanic T, Tolaney SM, Turner NC, Curigliano G, Loibl S, Paluch-Shimon S, Harbeck N; ESMO Guidelines Committee. Electronic address: clinicalguidelines@esmo.org. ESMO Clinical Practice Guideline for the diagnosis, staging and treatment of patients with metastatic breast cancer. Ann Oncol. 2021 Dec;32(12):1475-1495. doi: 10.1016/j.annonc.2021.09.019. Epub 2021 Oct 19. No abstract available. PMID 34678411
- [Background] Lowrance WT, Breau RH, Chou R, Chapin BF, Crispino T, Dreicer R, Jarrard DF, Kibel AS, Morgan TM, Morgans AK, Oh WK, Resnick MJ, Zietman AL, Cookson MS. Advanced Prostate Cancer: AUA/ASTRO/SUO Guideline PART II. J Urol. 2021 Jan;205(1):22-29. doi: 10.1097/JU.0000000000001376. Epub 2020 Sep 22. PMID 32960678
- [Background] Gonzalez Del Alba A, Mendez-Vidal MJ, Vazquez S, Castro E, Climent MA, Gallardo E, Gonzalez-Billalabeitia E, Lorente D, Maroto JP, Arranz JA. SEOM clinical guidelines for the treatment of advanced prostate cancer (2020). Clin Transl Oncol. 2021 May;23(5):969-979. doi: 10.1007/s12094-021-02561-5. Epub 2021 Feb 24. PMID 33625671
- [Background] Garvelink MM, Boland L, Klein K, Nguyen DV, Menear M, Bekker HL, Eden KB, LeBlanc A, O'Connor AM, Stacey D, Legare F. Decisional Conflict Scale Use over 20 Years: The Anniversary Review. Med Decis Making. 2019 May;39(4):301-314. doi: 10.1177/0272989X19851345. Epub 2019 May 29. PMID 31142194
- [Background] Lee YH, Chou XY, Lai YH, Liang YH, Hung CT, Hsaio CC, Gao ZX. Decisional conflict and its determinants among patients with cancer undergoing immunotherapy combined with chemotherapy or targeted therapy: a cross-sectional study. Sci Rep. 2023 Aug 5;13(1):12715. doi: 10.1038/s41598-023-39280-6. PMID 37543690
- [Background] van Steenhoven JEC, den Dekker BM, Kuijer A, van Diest PJ, Nieboer P, Zuetenhorst JM, Imholz ALT, Siesling S, van Dalen T. Patients' perceptions of 70-gene signature testing: commonly changing the initial inclination to undergo or forego chemotherapy and reducing decisional conflict. Breast Cancer Res Treat. 2020 Jul;182(1):107-115. doi: 10.1007/s10549-020-05683-6. Epub 2020 May 19. PMID 32430679
- [Background] Hoesseini A, Dorr MC, Dronkers EAC, de Jong RJB, Sewnaik A, Offerman MPJ. Decisional Conflict in Patients With Head and Neck Cancer. JAMA Otolaryngol Head Neck Surg. 2023 Feb 1;149(2):160-167. doi: 10.1001/jamaoto.2022.4269. PMID 36547952
- [Background] Ribi K, Kalbermatten N, Eicher M, Strasser F. Towards a novel approach guiding the decision-making process for anticancer treatment in patients with advanced cancer: framework for systemic anticancer treatment with palliative intent. ESMO Open. 2022 Jun;7(3):100496. doi: 10.1016/j.esmoop.2022.100496. Epub 2022 May 18. PMID 35597176
- [Background] Fondo Colombiano de Enfermedades de Alto Costo. Situación del cáncer en la población adulta atendida en el SGSSS de Colombia 2022. Bogotá: Cuenta de Alto Costo (CAC); 2023. 58 p.
- [Background] Ferlay J, Bray F, Soerjomataram I, Znaor A, Ervik M, Lam F, et al. International Agency for Research on Cancer. 2024 (cited 2024 Sep 7). Global Cancer Observatory: Cancer Today.
- [Background] Saini KS, Twelves C. Determining lines of therapy in patients with solid cancers: a proposed new systematic and comprehensive framework. Br J Cancer. 2021 Jul;125(2):155-163. doi: 10.1038/s41416-021-01319-8. Epub 2021 Apr 13. PMID 33850304